CLINICAL TRIAL: NCT04224272
Title: Phase 2a Study of ZW25 in Combination With Palbociclib Plus Fulvestrant
Brief Title: A Study of ZW25 (Zanidatamab) With Palbociclib Plus Fulvestrant in Patients With HER2+/HR+ Advanced Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Jazz Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ZWI-ZW25-202; 2019-002956-18 (EudraCT Number)
Expanded Access: NCT04578444 (No longer available)
Record Dates: First submitted 2020-01-07; First posted 2020-01-13 (Actual); Results first posted 2024-08-14 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: HER2+/HR+ Breast Cancer
Keywords: HER2; HR; Bispecific antibody; Biparatopic antibody; Immunotherapy; Breast cancer; Chemotherapy; Palbociclib; Fulvestrant
MeSH Terms: conditions — Breast Neoplasms | interventions — zanidatamab; palbociclib; Fulvestrant

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- ZW25 (zanidatamab) + palbociclib + fulvestrant (Experimental): ZW25 (zanidatamab) plus palbociclib, fulvestrant
  Interventions: Drug: ZW25 (Zanidatamab); Drug: Palbociclib; Drug: Fulvestrant

INTERVENTIONS:
Drug: ZW25 (Zanidatamab) — Administered intravenously
Drug: Palbociclib — Administered orally
Drug: Fulvestrant — Administered as an intramuscular injection

SUMMARY:
This is a multicenter, Phase 2a, open-label, 2-part study to investigate the safety, tolerability, and anti-tumor activity of ZW25 (zanidatamab) in combination with palbociclib plus fulvestrant. Eligible patients include those with locally advanced (unresectable) and/or metastatic human epidermal growth factor receptor 2 (HER2)-positive, hormone receptor (HR)-positive breast cancer.

DETAILED DESCRIPTION:
Part 1 of the study will first evaluate the safety and tolerability of ZW25 in combination with palbociclib plus fulvestrant and will confirm the recommended doses (RDs) of ZW25 and palbociclib in this combination. Part 2 of the study will evaluate the anti-tumor activity of the combination of ZW25 with palbociclib plus fulvestrant at the RD level in patients with HER2-positive, HR-positive advanced breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically-confirmed diagnosis of breast cancer with evidence of locally advanced (unresectable) and/or metastatic disease. All patients in both Parts 1 and 2 must have HER2-positive and HR-positive disease.
* Received prior treatment with trastuzumab, pertuzumab, AND ado-trastuzumab emtansine (T-DM1); disease progression during or after the most recent prior therapy. Patients in any part of the study who did not receive pertuzumab or T-DM1 because of lack of access (e.g., due to insurance coverage or because they were treated prior to regulatory agency approval of the agent in a relevant indication) or due to medical ineligibility for treatment with T-DM1 (e.g., history of severe infusion reactions to trastuzumab, >/= Grade 2 peripheral neuropathy, or platelet count < 100 x 10^9/L) may be eligible for the study. Prior treatment with endocrine therapy in the neoadjuvant, adjuvant, and/or metastatic setting is permitted.
* Sites of disease assessible per RECIST version 1.1 (both measurable and non-measurable disease allowed)
* An Eastern Cooperative Oncology Group (ECOG) Performance Status score of 0 or 1
* Adequate organ function
* Adequate cardiac left ventricular function, as defined by left ventricular ejection fraction (LVEF) >/= institutional standard of normal

Exclusion Criteria:

* Prior treatment with trastuzumab, pertuzumab, lapatinib, T-DM1, or other anti-HER2-targeted therapy </= 3 weeks before the first dose of ZW25
* Prior treatment with chemotherapy, other anti-cancer therapy not otherwise specified, or hormonal cancer therapy </= 3 weeks before the first dose of ZW25
* Prior treatment with palbociclib or any other CDK4/6 inhibitor, including experimental agents
* History of myocardial infarction or unstable angina within 6 months prior to enrollment, troponin levels consistent with myocardial infarction, or clinically significant cardiac disease, such as ventricular arrhythmia requiring therapy, uncontrolled hypertension, or any history of symptomatic congestive heart failure (CHF)
* QTc Fridericia (QTcF) > 470 ms
* Grade 2 or greater pneumonitis and/or interstitial lung disease, including pulmonary fibrosis, or other clinically significant infiltrative pulmonary disease not related to lung metastases
* Active hepatitis B or hepatitis C infection
* Acute or chronic uncontrolled renal disease, pancreatitis, or severe liver disease (Child-Pugh Class C)
* Known infection with Human Immunodeficiency Virus (HIV)-1 or HIV-2 (Exception: patients with well controlled-HIV [e.g., cluster of differentiation 4 (CD4)-positive T-cell count > 350 mm3 and undetectable viral load] are eligible.)
* Prior or concurrent malignancy whose natural history or treatment has the potential to interfere with the safety or efficacy assessment of the investigational regimen
* Brain metastases: Untreated central nervous system (CNS) metastases, symptomatic CNS metastases, or radiation treatment for CNS metastases within 4 weeks of start of study treatment. Stable, treated brain metastases are allowed (defined as patients who are off steroids and anticonvulsants and are neurologically stable for at least 1 month at the time of screening).
* History of or ongoing leptomeningeal disease
* Grade 3 or greater peripheral neuropathy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2020-06-10 (Actual); Primary Completion 2023-04-28 (Actual); Study Completion 2025-06-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (13):
- United States (3):
  - UCLA Hematology/Oncology Parkside, Santa Monica, California
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - Seattle Cancer Care Alliance, Seattle, Washington
- Canada (4):
  - Tom Baker Cancer Centre, Calgary, Alberta
  - The Ottawa Hospital Cancer Centre, Ottawa, Ontario
  - Sunnybrook Research Institute, Toronto, Ontario
  - Jewish General Hospital, Montreal, Quebec
- Spain (6):
  - Hospital General Universitario de Elche, Elche, Alicante
  - Hospital Universitario Vall d'Hebrón, Barcelona
  - Hospital Ruber Internacional, Madrid
  - Hospital Universitario Virgen de la Victoria, Málaga
  - Hospital Universitario Virgen del Rocío, Seville
  - Hospital Clínico Universitario de Valencia, Valencia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Escriva-de-Romani S, Cejalvo JM, Alba E, Friedmann J, Rodriguez-Lescure A, Savard MF, Pezo RC, Gion M, Ruiz-Borrego M, Hamilton E, Pluard T, Webster M, Beeram M, Linden H, Saura C, Shpektor D, Salim B, Harvey P, Hurvitz SA. Zanidatamab plus palbociclib and fulvestrant in previously treated patients with hormone receptor-positive, HER2-positive metastatic breast cancer: primary results from a two-part, multicentre, single-arm, phase 2a study. Lancet Oncol. 2025 Jun;26(6):745-758. doi: 10.1016/S1470-2045(25)00140-8. Epub 2025 May 5. PMID 40339592

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 51 participants who met all eligibility criteria were enrolled and received treatment.
Groups:
- ZW25 (Zanidatamab) + Palbociclib + Fulvestrant: Participants who received an intravenous dose of 20 mg/kg ZW25 (zanidatamab) every 2 weeks (Q2W) in combination with an oral administration of 125 mg palbociclib once daily from Days 1 to 21, and an intramuscular injection of 500 mg fulvestrant Q2W for 3 doses (Cycle 1 Days 1 and 15 and Cycle 2 Day 1), and every 4 weeks (Q4W) thereafter.
Period: Part 1 - Dose Finding
Arm/Group | ZW25 (Zanidatamab) + Palbociclib + Fulvestrant
Started | 8
Completed | 1
Not Completed | 7
Not completed — Death | 4
Not completed — Withdrawal by Subject | 2
Not completed — Lost to Follow-up | 1
Period: Part 2 - Dose Expansion
Arm/Group | ZW25 (Zanidatamab) + Palbociclib + Fulvestrant
Started | 43
Completed | 30
Not Completed | 13
Not completed — Death | 10
Not completed — Withdrawal by Subject | 3

BASELINE CHARACTERISTICS:
Population: The baseline demographic characteristics were assessed in the Safety Analysis Set.
Groups:
- ZW25 (Zanidatamab) + Palbociclib + Fulvestrant: Participants who received intravenous dose of 20 mg/kg ZW25 (zanidatamab) every 2 weeks (Q2W) in combination with an oral administration of 125 mg palbociclib once daily from Days 1 to 21, and an intramuscular injection of 500 mg fulvestrant Q2W for 3 doses (Cycle 1 Days 1 and 15 and Cycle 2 Day 1), and every 4 weeks (Q4W) thereafter.
Arm/Group | ZW25 (Zanidatamab) + Palbociclib + Fulvestrant
Number analyzed (Participants) | 51
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.7 (10.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 49
  Male | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 2
  Black or African American | 1
  White | 42
  Multiple | 1
  Other | 1
  Unknown | 3
  Not Reported | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dose-Limiting Toxicities
Description: Dose-limiting toxicities, defined using NCI CTCAE version 5.0, are events that 1) occur following administration of ZW25, palbociclib, and fulvestrant, or any combination of ZW25 and 1 or more of these drugs; and 2) meet the criteria as specified in the protocol.
Time Frame: Cycle 1 Day 1 to Day 28 (each cycle is 28 days)
Population: Dose-limiting toxicities were assessed in participants with available data in the Safety Analysis Set.
Measure: Count of Participants; unit: Participants
Arm/Group | ZW25 (Zanidatamab) + Palbociclib + Fulvestrant
Number analyzed (Participants) | 8
Participants | 1

2. Secondary Outcome: Number of Participants Reporting Any Treatment-emergent Adverse Event, Serious Adverse Event, and Adverse Event of Special Interest
Description: A treatment-emergent adverse events (TEAEs) was defined as an adverse event (AE) with onset on or after 1st dose of study treatment through 30 days after final dose of study treatment inclusive. An AE is classified as a serious adverse event (SAE) if fatal, life threatening, requires hospitalization, is disabling/incapacitating, causes congenital anomaly or birth defect, and medically significant. Adverse events of special interest (AESI) include absolute decreases in LVEF greater than or equal to 10 percentage points from baseline, symptomatic heart failure, infusion-related reactions, and all greater than or equal to Grade 2 events of pneumonitis and/or interstitial lung disease, including pulmonary fibrosis.
Time Frame: From the start of dosing of any study drug up until 30 days after last study dose, up to approximately 2 years 10 months
Population: Safety data were assessed in the Safety Analysis Set.
Measure: Count of Participants; unit: Participants
Arm/Group | ZW25 (Zanidatamab) + Palbociclib + Fulvestrant
Number analyzed (Participants) | 51
Participants
  TEAE | 51
  SAE | 8
  AESI | 10

3. Primary Outcome: Number of Participants Reporting Grade 3 or Higher Treatment-emergent Adverse Events
Description: A treatment-emergent adverse event occurs after the start of study treatment and is defined as any unfavorable or unintended symptom, sign, or disease (including abnormal lab) temporally associated with the use of treatment that may or may not be considered related to treatment. TEAEs were coded using MedDRA v24.0.
Time Frame: Baseline from the start of dosing of any study drug up until 30 days after last study dose, up to approximately 2 years 10 months.
Population: Treatment-emergent adverse events were assessed in the Safety Analysis Set.
Measure: Count of Participants; unit: Participants
Arm/Group | ZW25 (Zanidatamab) + Palbociclib + Fulvestrant
Number analyzed (Participants) | 51
Participants
  Any Blood and Lymphatic System Disorders AE | 20
  Neutropenia | 16
  Anaemia | 6
  Thrombocytopenia | 3
  Any Gastrointestinal Disorder AE | 13
  Diarrhoea | 8
  Abdominal pain | 1
  Duodenal ulcer | 1
  Gastric ulcer | 1
  Nausea | 1
  Small intestinal obstruction | 1
  Stomatitis | 1
  Vomiting | 1
  Any Investigation AE | 12
  Neutrophil count decreased | 11
  Ejection fraction decreased | 1
  Transaminases increased | 1
  White blood cell count decreased | 1
  Any Metabolism and Nutrition Disorder AE | 8
  Hypokalaemia | 4
  Hypomagnesaemia | 3
  Hypercalcaemia | 2
  Any General Disorders and Administration Site Conditions AE | 2
  Fatigue | 1
  Pyrexia | 1
  Any Infections and Infestations AE | 2
  COVID-19 pneumonia | 1
  Psoas abscess | 1
  Staphylococcal bacteraemia | 1
  Any Respiratory, Thoracic and Mediastinal Disorder AE | 2
  Pleural effusion | 1
  Pneumothorax | 1
  Any Renal and Urinary Disorder AE | 1
  Acute kidney injury | 1
  Any Skin and Subcutaneous Tissue Disorder AE | 1
  Rash maculo-papular | 1

4. Primary Outcome: Progression-free Survival 6
Description: The progression-free survival at 6 months (PFS6) is a binary endpoint variable based on the progression-free survival (PFS) time, defined as the proportion of participants having PFS time greater than or equal to 24 weeks (168 days).
Time Frame: 6 months from first dose of any study drug to the date of documented disease progression or death
Population: Progression-free survival 6 will be assessed in the Safety Analysis Set.
Measure: Count of Participants; unit: Participants
Arm/Group | ZW25 (Zanidatamab) + Palbociclib + Fulvestrant
Number analyzed (Participants) | 51
Participants | 34

5. Secondary Outcome: Maximum Serum Concentration of ZW25
Time Frame: Cycle 1, Days 1, 2, 5, 15; Cycle 2, Days 1 and 15; Day 1 of all subsequent cycles (each cycle is 28 days); and end of treatment, up to approximately 5 years 4 months
Reporting Status: Not Posted, anticipated posting 2026-10

6. Secondary Outcome: Trough Concentration of ZW25
Time Frame: as for outcome 5
Reporting Status: Not Posted, anticipated posting 2026-10

7. Secondary Outcome: Incidence of Anti-drug Antibodies (ADAs)
Time Frame: Cycles 1 and 2, Day 15; Day 1 of all subsequent cycles (each cycle is 28 days); end of treatment, 30 days post-last dose (safety follow up), and every 8 weeks (efficacy follow up), up to approximately 5 years 4 months
Reporting Status: Not Posted, anticipated posting 2026-10

8. Secondary Outcome: Objective Response Rate
Time Frame: Baseline up to end of study, approximately 5 years 4 months
Reporting Status: Not Posted, anticipated posting 2026-10

9. Secondary Outcome: Duration of Response
Time Frame: Baseline up to end of study, approximately 5 years 4 months
Reporting Status: Not Posted, anticipated posting 2026-10

10. Secondary Outcome: Disease Control Rate
Time Frame: Baseline up to end of study, approximately 5 years 4 months
Reporting Status: Not Posted, anticipated posting 2026-10

11. Secondary Outcome: Progression-free Survival
Time Frame: Baseline up to end of study, approximately 5 years 4 months
Reporting Status: Not Posted, anticipated posting 2026-10

12. Secondary Outcome: Overall Survival
Time Frame: Baseline up to end of study, approximately 5 years 4 months
Reporting Status: Not Posted, anticipated posting 2026-10

13. Secondary Outcome: Incidence of Lab Abnormalities
Time Frame: Baseline up to end of study, approximately 5 years 4 months
Reporting Status: Not Posted, anticipated posting 2026-10

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the start of dosing of any study drug up until 30 days after last study dose, up to approximately 2 years 10 months.
Arm/Group | ZW25 (Zanidatamab) + Palbociclib + Fulvestrant
All-Cause Mortality (participants affected / at risk) | 14/51
Serious Adverse Events (participants affected / at risk) | 8/51
Other Adverse Events (participants affected / at risk) | 51/51
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ZW25 (Zanidatamab) + Palbociclib + Fulvestrant (N=51)
Duodenal ulcer (Gastrointestinal disorders) | 1
Gastric ulcer (Gastrointestinal disorders) | 1
Small intestinal obstruction (Gastrointestinal disorders) | 1
COVID-19 (Infections and infestations) | 1
COVID-19 pneumonia (Infections and infestations) | 1
Psoas abscess (Infections and infestations) | 1
Staphylococcal bacteraemia (Infections and infestations) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1
Anaemia (Blood and lymphatic system disorders) | 1
Transaminases increased (Investigations) | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 1
Acute kidney injury (Renal and urinary disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | ZW25 (Zanidatamab) + Palbociclib + Fulvestrant (N=51)
Diarrhoea (Gastrointestinal disorders) | 47
Nausea (Gastrointestinal disorders) | 27
Stomatitis (Gastrointestinal disorders) | 21
Vomiting (Gastrointestinal disorders) | 17
Abdominal pain (Gastrointestinal disorders) | 11
Dyspepsia (Gastrointestinal disorders) | 8
Constipation (Gastrointestinal disorders) | 5
Abdominal pain upper (Gastrointestinal disorders) | 4
Abdominal distension (Gastrointestinal disorders) | 3
Asthenia (General disorders) | 19
Fatigue (General disorders) | 10
Pyrexia (General disorders) | 5
Injection site pain (General disorders) | 3
Neutropenia (Blood and lymphatic system disorders) | 19
Anaemia (Blood and lymphatic system disorders) | 16
Thrombocytopenia (Blood and lymphatic system disorders) | 8
COVID-19 (Infections and infestations) | 10
Urinary tract infection (Infections and infestations) | 9
Nasopharyngitis (Infections and infestations) | 4
Decreased appetite (Metabolism and nutrition disorders) | 12
Hypokalaemia (Metabolism and nutrition disorders) | 10
Hypomagnesaemia (Metabolism and nutrition disorders) | 7
Neutrophil count decreased (Investigations) | 14
Ejection fraction decreased (Investigations) | 8
Platelet count decreased (Infections and infestations) | 7
Weight decreased (Investigations) | 6
White blood cell count decreased (Investigations) | 4
Blood alkaline phosphatase increased (Investigations) | 3
Rash (Skin and subcutaneous tissue disorders) | 9
Pruritus (Skin and subcutaneous tissue disorders) | 5
Alopecia (Skin and subcutaneous tissue disorders) | 4
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 4
Dry skin (Skin and subcutaneous tissue disorders) | 3
Muscle spasms (Musculoskeletal and connective tissue disorders) | 9
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5
Arthralgia (Musculoskeletal and connective tissue disorders) | 4
Back pain (Musculoskeletal and connective tissue disorders) | 4
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 3
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 10
Cough (Respiratory, thoracic and mediastinal disorders) | 5
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3
Headache (Nervous system disorders) | 9
Dizziness (Nervous system disorders) | 5
Paraesthesia (Nervous system disorders) | 4
Peripheral sensory neuropathy (Nervous system disorders) | 3
Insomnia (Psychiatric disorders) | 3
Hot flush (Vascular disorders) | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-09-26): https://cdn.clinicaltrials.gov/large-docs/72/NCT04224272/Prot_SAP_000.pdf